CLINICAL TRIAL: NCT03238196
Title: A Phase Ib Trial of Fulvestrant, Palbociclib (CDK4/6 Inhibitor) and Erdafitinib (JNJ- 42756493,Pan-FGFR Tyrosine Kinase Inhibitor) in ER+/HER2-/FGFR-Amplified Metastatic Breast Cancer (MBC)
Brief Title: Fulvestrant, Palbociclib and Erdafitinib in ER+/HER2-/FGFR-amplified Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brent Rexer, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VICC BRE 16126
Record Dates: First submitted 2017-07-24; First posted 2017-08-03 (Actual); Results first posted 2023-02-16 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Breast Cancer
Keywords: FGFR inhibitor; ER+ metastatic breast cancer; CDK4/6 inhibitor; Endocrine therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — erdafitinib; palbociclib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Escalation (Experimental): Fulvestrant - injection into muscle 1 time per month
  Palbociclib capsule taken by mouth 1 time per day every 21 days followed by 1 week of rest (no drug taken)
  Erdafitinib tablet taken by mouth 1 time per day
  Interventions: Drug: Erdafitinib; Drug: Palbociclib; Drug: Fulvestrant
- Expansion (Experimental): Fulvestrant - injection into muscle 1 time per month
  Palbociclib capsule taken by mouth 1 time per day every 21 days followed by 1 week of rest (no drug taken)
  Erdafitinib tablet taken by mouth 1 time per day
  Interventions: Drug: Erdafitinib; Drug: Palbociclib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Erdafitinib — 4mg - 8mg
  Other Names: JNJ-42756493
Drug: Palbociclib — 125 mg
  Other Names: Ibrance
Drug: Fulvestrant — 500 mg
  Other Names: Faslodex

SUMMARY:
This is an open-label, multi-institution, phase Ib trial that evaluates the safety and tolerability and preliminary anti-tumor activity of fulvestrant, palbociclib and erdafitinib in patients with ER+/HER2-/FGFR-amplified metastatic breast cancer.

DETAILED DESCRIPTION:
Primary Objectives

To determine the safety and tolerability of fulvestrant, palbociclib and erdafitinib in patients with ER+/HER2-/FGFR-amplified MBC.

Secondary Objectives

* To determine the anti-tumor effect of fulvestrant, palbociclib and erdafitinib in patients with ER+/HER2-/FGFR-amplified MBC.
* Pharmacokinetic assessments of erdafitinib

Correlative Objectives

* To determine the therapeutic predictive role of FGFR1-4, CCND1-2, CDK4 and CDK6 amplifications, and RB1 and ESR1 mutations on clinical outcome
* To determine if the FGFR1 amplification levels is an early surrogate of response
* To determine if the cfDNA results at disease progression show new genomic alterations potentially associated with resistance to CDK4/6 and FGFR inhibition
* To determine pharmacodynamic biomarkers of FGFR inhibition

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to swallow and retain oral medication
* Patients must be ≥ 18 years of age
* Female patients of no childbearing potential must be post-menopausal. Postmenopausal female subjects should be defined prior to protocol enrollment by any of the following:
* Participants at least 60 years of age; OR
* Participants under 60 years of age and naturally (spontaneous, no alternative pathologic or physiological cause) amenorrhea for at least 12 months; OR
* Medical ovarian failure confirmed by follicle-stimulating hormone (FSH) and estradiol levels in the post menopausal range per local institutional normal range; OR
* Prior bilateral oophorectomy; OR
* Prior radiation castration with amenorrhea for at least 6 months; OR
* Treatment with a luteinizing hormone-releasing hormone (LH-RH) agonist (such as goserelin acetate or leuprolide acetate) is permitted for induction of ovarian suppression as long as it has been initiated at least 28 days prior to study enrollment
* Patients must have ECOG performance status 0 - 1
* Patients must have clinical stage IV or inoperable locoregional recurrent invasive mammary carcinoma that is:
* ER+ and/or PgR+ (≥ 1% positive stained cells) by immunohistochemistry (IHC)
* HER2-negative (by IHC or FISH, per ASCO guidelines)
* FGFR1 - 4 amplified
* Patients must have evaluable (may have either measurable or non-measurable) disease
* Patients must have available tissue for FGFR determination
* Patients must have had at least one line of therapy in the metastatic setting
* Current use of any of the drugs listed on the Cautionary Concomitant Med list has to be approved by the Study Chair
* Patients must have adequate hematologic, hepatic and renal function. All laboratory tests must be obtained within 2 weeks from study drug initiation. These include:
* ANC ≥ 1,500/mm3
* Platelet count ≥ 100,000/mm3
* HgB ≥ 9.0 g/dL
* Creatinine clearance ≥ 40 mL/min/1.73 m2
* SGOT, SGPT ≤ 2.5 x ULN if no liver metastasis present; SGOT, SGPT ≤ 4 x ULN if liver metastasis present
* Albumin ≥ 2.0 g/dL
* Total serum bilirubin ≤ 1.5 x ULN (≤ 3 x ULN or direct bilirubin ≤ 1.5 x ULN if known Gilbert's syndrome)
* Potassium within institutional normal limits
* Phosphorus ≤ institutional upper limit of normal

Exclusion Criteria:

* Prior use of an FGFR inhibitor
* More than 2 lines of chemotherapy in the metastatic setting. No limit on endocrine therapy lines. Prior exposure to CDK4/6 inhibitor acceptable.
* Radiation therapy ≤ 2 weeks prior to study entry. Patients who have received prior radiotherapy must have recovered from toxicity (≤ grade 1) induced by this treatment (except for alopecia)
* Prior cancer therapy (except for endocrine therapy) must have been discontinued for 1 week prior to initiation of study drugs
* Concurrent anti-cancer therapy other than the ones specified in the protocol is not permitted during study participation. Bisphosphonates or denosumab are allowed
* Major surgery within 4 weeks of enrollment
* Herbal preparations are not allowed throughout the study, and should be discontinued 14 days prior to initiation of study treatment
* Any corneal or retinal abnormality likely to increase the risk of eye toxicity, such as:
* Current corneal pathology such as keratitis, keratoconjunctivitis, keratopathy, corneal abrasion, inflammation or ulceration
* Uncontrolled glaucoma despite standard of care therapy
* Diabetic retinopathy with macular edema
* Known active wet, age-related macular degeneration (AMD)
* Known central serous retinopathy (CSR) or retinal vascular occlusion (RVO)
* Uncontrolled intercurrent illness including, but not limited to:
* Malabsorption syndrome significantly affecting gastrointestinal function
* Ongoing or active infection requiring antibiotics/antivirals
* Impairment of lung function (COPD > grade 2, lung conditions requiring oxygen therapy)
* Symptomatic congestive heart failure
* Unstable angina pectoris, angioplasty, stenting, or myocardial infarction within 6 months
* Clinically significant cardiac arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia that is symptomatic or requires treatment [National Cancer Institute -Common Terminology Criteria for Adverse Events, Version 4.03, grade 3]
* QTcF ≥ 480 msec on screening EKG
* Known history of clinically significant QT/QTc prolongation or Torsades de Pointes(TdP)
* ST depression or elevation of ≥ 1.5 mm in 2 or more leads
* Diarrhea of any cause ≥ CTCAE grade 2 that does not resolve within a few days when adequately treated with anti-diarrhea medications
* Psychiatric illness/social situations that would compromise patient safety or limit compliance with study requirements including maintenance of a compliance/pill diary
* Symptomatic brain metastases (patients with a history of brain metastases must be clinically stable for more than 4 weeks from completion of radiation treatment and be off steroids)
* Known history of chronic liver or chronic renal failure
* Poor wound healing capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2024-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brent Rexer, MD, PhD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (6):
- United States (6):
  - University of Alabama, Birmingham, Alabama
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baptist Memorial Hospital MEMPHIS, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Southwestern Simmons Comprehensive Cancer Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Ericsson PI, Unni N, Jhaveri K, Stringer-Reasor E, Liu Q, Wang Y, Sanchez V, Garcia G, Sanders ME, Lehmann BD, Balko JM, Park B, Rexer BN, Mayer IA, Arteaga CL. Phase Ib Trial of Fulvestrant, Palbociclib, and Erdafitinib, a pan-FGFR Tyrosine Kinase Inhibitor, in HR+/HER2- Metastatic Breast Cancer. Clin Cancer Res. 2025 Sep 2;31(17):3652-3661. doi: 10.1158/1078-0432.CCR-24-3803. PMID 40627530
- See also: Clinical Trials Webpage - Vanderbilt-Ingram Cancer Center — http://www.vicc.org/ct/protocols.php?cancer-type=Breast
- See also: Mycancergenome - FGFR1 Webpage — https://www.mycancergenome.org/content/disease/breast-cancer/fgfr1/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited to this trial from August 2017 to January 2021 at five medical centers.
Groups:
- Expansion: Fulvestrant - injection into muscle 1 time per month
  Palbociclib capsule taken by mouth 1 time per day every 21 days followed by 1 week of rest (no drug taken)
  Erdafitinib tablet taken by mouth 1 time per day
  Erdafitinib: 6 mg
  Palbociclib: 125 mg
  Fulvestrant: 500 mg
- Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 5mg (Escalation): Participants who were treated with Fulvestrant 500mg, Palbociclib 125mg and Erdafitinib 5mg.
- Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 6mg (Escalation): Participants who were treated with Fulvestrant 500mg, Palbociclib 125mg and Erdafitinib 6mg.
- Fulvestrant 500mg, Palbociclib 125mg and Erdafitinib 8mg (Escalation): Participants who were treated with Fulvestrant 500mg, Palbociclib 125mg and Erdafitinib 8mg.
Period: Overall Study
Arm/Group | Expansion | Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 5mg (Escalation) | Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 6mg (Escalation) | Fulvestrant 500mg, Palbociclib 125mg and Erdafitinib 8mg (Escalation)
Started | 22 | 3 | 6 | 4
Completed | 0 | 0 | 0 | 0
Not Completed | 22 | 3 | 6 | 4
Not completed — Adverse Event | 3 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 4 | 1 | 1 | 0
Not completed — Disease progression | 14 | 2 | 3 | 2
Not completed — Still on treatment | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Expansion: Fulvestrant - injection into muscle 1 time per month
  Palbociclib capsule taken by mouth 1 time per day every 21 days followed by 1 week of rest (no drug taken)
  Erdafitinib tablet taken by mouth 1 time per day
  Erdafitinib: 6mg
  Palbociclib: 125 mg
  Fulvestrant: 500 mg
- Total: Total of all reporting groups
Arm/Group | Expansion | Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 5mg (Escalation) | Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 6mg (Escalation) | Fulvestrant 500mg, Palbociclib 125mg and Erdafitinib 8mg (Escalation) | Total
Number analyzed (Participants) | 22 | 3 | 6 | 4 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 2 | 5 | 3 | 28
  >=65 years | 4 | 1 | 1 | 1 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 3 | 6 | 4 | 35
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 14 | 3 | 3 | 1 | 21
  Unknown or Not Reported | 7 | 0 | 3 | 3 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2
  White | 17 | 2 | 3 | 2 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 22 | 3 | 6 | 4 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT) in the First Cycle for the Determination of the Maximum Tolerated Dose (MTD)
Description: Number of participants with DLT in the first cycle for the determination of the MTD.
Time Frame: From the time of randomization up to 4 weeks of treatment (cycle 1), for each patient
Population: Participants who were treated with Fulvestrant 500mg, Palbociclib 125mg and Erdafitinib in Escalation phase.
Measure: Number; unit: participants
Groups:
- Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 5mg (Escalation): Participants take Erdafitinib 5mg orally once a day in 28-day cycle, with Fulvestrant 500mg IM once every 28 days (for cycle 1 it is administered at day 15) and Palbociclib 125mg daily for 21 days out of a 28-day cycle.
- Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 6mg (Escalation): Participants take Erdafitinib 6mg orally once a day in 28-day cycle, with Fulvestrant 500mg IM once every 28 days (for cycle 1 it is administered at day 15) and Palbociclib 125mg daily for 21 days out of a 28-day cycle.
- Fulvestrant 500mg, Palbociclib 125mg and Erdafitinib 8mg (Escalation): Participants take Erdafitinib 8mg orally once a day in 28-day cycle, with Fulvestrant 500mg IM once every 28 days (for cycle 1 it is administered at day 15) and Palbociclib 125mg daily for 21 days out of a 28-day cycle.
Arm/Group | Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 5mg (Escalation) | Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 6mg (Escalation) | Fulvestrant 500mg, Palbociclib 125mg and Erdafitinib 8mg (Escalation)
Number analyzed (Participants) | 3 | 6 | 4
participants | 0 | 0 | 2

2. Secondary Outcome: Progression-free Survival
Description: Assessment of clinical impact [anti-tumor effect] of the combination of erdafitinib, palbociclib and fulvestrant in patients with ER+/ FGFR amplified metastatic breast cancer will be assessed by measuring the interval (in months) between treatment initiation and disease progression. Progression-free survival (PFS) time is defined as the time from treatment initiation to progression date or death (whichever comes first). Those alive without prpgression is censored at the last date of known alive. Median PFS time and 95% confidence intervals are obtained using Kaplan-meier method.
Time Frame: Imaging studies will be performed every 8 weeks from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
Population: All participants. This study was a single-arm dose escalation/dose expansion study. Therefore we did not subdivide the dose level groups for the secondary outcomes as the study was not powered for any intra-arm comparisons of clinical benefit.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Escalation and Expansion: Fulvestrant - injection into muscle 1 time per month
  Palbociclib capsule taken by mouth 1 time per day every 21 days followed by 1 week of rest (no drug taken)
  Erdafitinib tablet taken by mouth 1 time per day
  Erdafitinib: 4mg - 8mg
  Palbociclib: 125 mg
  Fulvestrant: 500 mg
Arm/Group | Escalation and Expansion
Number analyzed (Participants) | 35
weeks | 12.4 [8.1 to 22.0]

3. Secondary Outcome: Overall Response Rate
Description: Assessment of clinical impact [anti-tumor effect] of the combination of erdafitinib, palbociclib and fulvestrant in patients with ER+/ FGFR amplified metastatic breast cancer by measure the rate (%) of complete and partial responses seen in patients with measurable disease. The response of a patient will be evaluated using Solid Tumor Response Criteria RECIST v1.1.
Time Frame: as for outcome 2
Population: Patients received the treatment and had valuable response data. This study was a single-arm dose escalation/dose expansion study. Therefore we did not subdivide the dose level groups for the secondary outcomes as the study was not powered for any intra-arm comparisons of clinical benefit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Escalation and Expansion
Number analyzed (Participants) | 31
percentage of participants | 9.7 [3.3 to 24.9]

4. Secondary Outcome: Clinical Benefit Rate (CBR; Complete Response + Partial Response + Stable Disease Without Disease Progression at 6 Months)
Description: Assessment of clinical impact [anti-tumor effect] of the combination of erdafitinib, palbociclib and fulvestrant in patients with ER+/ FGFR amplified metastatic breast cancer by measure the rate (%) of complete and partial responses + stability of disease at 6 months seen in patients with measurable disease. Response of a patient was evaluated using Solid Tumor Response Criteria -RECIST v1.1.
Time Frame: From the time of randomization up to 6 months for each patient
Population: Participants received the treatment and had evaluable response data. This study was a single-arm dose escalation/dose expansion study. Therefore we did not subdivide the dose level groups for the secondary outcomes as the study was not powered for any intra-arm comparisons of clinical benefit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Escalation and Expansion
Number analyzed (Participants) | 31
percentage of participants | 64.5 [46.9 to 78.9]

5. Secondary Outcome: Pharmacokinetic Assessment of Erdafitinib - Area Under the Curve (AUC)
Description: The area under the plasma concentration-time curve from time zero to the last measurable concentration
Time Frame: From the time of randomization up to 4 weeks of treatment for each patient
Population: Patients who actually received erdafitinib 5m, 6 mg and 8mg and participated the PK study by measuring the blood plasma concentration. One patients could have PK data at different cycles and days.
  For dose 5mg, 7 patients had 14 PK data. For daose 6mg, 6 patients had 11 PK data. For dose8mg, 4 patients had 8 PK data.
Measure: Mean (Standard Deviation); unit: ng/ml.hr
Arm/Group | Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 5mg (Escalation) | Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 6mg (Escalation) | Fulvestrant 500mg, Palbociclib 125mg and Erdafitinib 8mg (Escalation)
Number analyzed (Participants) | 7 | 6 | 4
ng/ml.hr | 1128 (608) | 718 (521) | 1268 (827)

6. Secondary Outcome: Pharmacokinetic Assessment of Erdafitinib - Cmax (Maximum Plasma Concentration)
Description: The maximum (peak) observed plasma drug concentration after oral dose administration
Time Frame: From the time of randomization up to 4 weeks of treatment for each patient
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 5mg (Escalation) | Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 6mg (Escalation) | Fulvestrant 500mg, Palbociclib 125mg and Erdafitinib 8mg (Escalation)
Number analyzed (Participants) | 7 | 6 | 8
ng/ml | 875 (625) | 668 (528) | 737 (348)

7. Secondary Outcome: Pharmacokinetic Assessment of Erdafitinib - Tmax
Description: Time to reach maximum (Cmax) plasma drug concentration after oral dose administration (time)
Time Frame: From the time of randomization up to 4 weeks of treatment for each patient
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 5mg (Escalation) | Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 6mg (Escalation) | Fulvestrant 500mg, Palbociclib 125mg and Erdafitinib 8mg (Escalation)
Number analyzed (Participants) | 7 | 6 | 4
hour | 2.8 (2.5) | 2.5 (1.8) | 2.8 (2.5)

8. Secondary Outcome: Pharmacokinetic Assessment of Erdafitinib - CL/F
Description: Apparent total body clearance of drug from the plasma after oral administration
Time Frame: From the time of randomization up to 4 weeks of treatment for each patient
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: l/hr
Arm/Group | Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 5mg (Escalation) | Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 6mg (Escalation) | Fulvestrant 500mg, Palbociclib 125mg and Erdafitinib 8mg (Escalation)
Number analyzed (Participants) | 7 | 6 | 4
l/hr | 5.5 (2.6) | 11.3 (5.5) | 8.6 (4.6)

9. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events [Tolerability]
Description: Assessment of adverse events throughout the study. The number of patients who had any grade of adverse events were reported.
Time Frame: From date of randomization until 28 days post treatment discontinuation from any cause, assessed up to 48 months
Population: All patients treated. This study was a single-arm dose escalation/dose expansion study. Therefore we did not subdivide the dose level groups for the secondary outcomes as the study was not powered for any intra-arm comparisons of clinical benefit.
Measure: Number; unit: patients
Groups:
- Escalation (6mg-8mg) and Expansion: Fulvestrant - injection into muscle 1 time per month
  Palbociclib capsule taken by mouth 1 time per day every 21 days followed by 1 week of rest (no drug taken)
  Erdafitinib tablet taken by mouth 1 time per day
  Erdafitinib: 6mg - 8mg
  Palbociclib: 125 mg
  Fulvestrant: 500 mg
Arm/Group | Escalation (6mg-8mg) and Expansion
Number analyzed (Participants) | 35
patients
  Oral mucositis, any grade | 27
  Hyperphosphatemia, any grade | 29
  Palmar-plantar erythrodysesthesia syndrome, any grade | 18
  Diarrhea, any grade | 14
  Constipation, any grade | 19
  Dysgeusia, any grade | 19
  Dry mouth, any grade | 18
  Nail alterations, any grade | 13
  Sore throat, any grade | 8
  Alopecia, any grade | 13
  Dry skin, any grade | 12
  Anorexia, any grade | 7
  Epistaxis, any grade | 9
  Dry eye, any grade | 10
  Skin ulceration, any grade | 2
  Vision changes/alterations, any grade | 6
  Neutrophil count decreased, grade 4 | 1
  Palmar-plantar erythrodysesthesia syndrome, grade 3 | 2
  Abdominal pain, any grade | 5
  Dizziness, any grade | 3
  Gastroesophageal reflux disease, any grade | 5
  Hypotension, any grade | 3
  Elevated ALT, any grade | 1
  Elevated AST, any grade | 3
  Colitis, any grade | 1
  Esophagitis, any grade | 2
  Eye keratopathy, any grade | 1
  Hyperkeratosis, any grade | 1
  Syncope, any grade | 1
  Neutropenia, any grade | 25
  Leucopenia, any grade | 15
  Anemia, any grade | 12
  Thrombocytopenia, any grade | 2
  Lymphopenia, any grade | 1
  Febrile neutropenia, any grade | 1
  Neutrophilia, any grade | 1
  Thromboembolic event, any grade | 1
  Fatigue, any grade | 15
  Nausea, any grade | 6
  Vomiting, any grade | 6

10. Other Pre Specified Outcome: Serial Measurements of Serum Phosphate, Calcium, Vitamin D, Parathyroid Hormone (PTH), FGF23, sFGFR2, sFGFR3, and sFGFR4
Description: Serial measurements of serum phosphate, calcium, vitamin D, PTH), FGF23, sFGFR2, sFGFR3, and sFGFR4 will be assessed to detect on target effects of FGFR inhibition (pharmacodynamic assessments).
Time Frame: During the first 8 weeks of treatment (days 1, 8, 15, 22 of cycle 1 and days 1 and 15 of cycle 2)
Reporting Status: Not Posted

11. Other Pre Specified Outcome: FGFR1 Amplification Levels by FISH and cfDNA
Description: The level of FGFR1 amplification assessed in tumors by fluorescence in situ hybridization (FISH) will be correlated with clinical outcome.
Time Frame: At study entry (baseline)
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Next Generation Sequencing
Description: Will determine if other genomic alterations other than FGFR amplifications correlate with clinical outcome.
Time Frame: At study entry (baseline)
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Plasma Cell-free Deoxyribonucleic Acid (cfDNA)
Description: Will determine if the cfDNA results at disease progression show new genomic alterations potentially associated with resistance to CDK4/6 and FGFR inhibition.
Time Frame: At study entry (baseline), at 4 weeks, and at study discontinuation from disease progression (for each patient), assessed up to 48 months.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Time frame for Serious adverse events and Other (Not Including Serious) Adverse Events: From time of informed consent signature to within 30 days of the last documented dose of study medication up to approximately 36 months.
Groups:
- Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 5mg: Participants who were treated with Fulvestrant 500mg, Palbociclib 125mg and Erdafitinib 5mg.
- Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 6mg: Participants who were treated with Fulvestrant 500mg, Palbociclib 125mg and Erdafitinib 6mg.
- Fulvestrant 500mg, Palbociclib 125mg and Erdafitinib 8mg: Participants who were treated with Fulvestrant 500mg, Palbociclib 125mg and Erdafitinib 8mg.
Arm/Group | Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 5mg | Expansion | Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 6mg | Fulvestrant 500mg, Palbociclib 125mg and Erdafitinib 8mg
All-Cause Mortality (participants affected / at risk) | 2/3 | 3/22 | 6/6 | 2/4
Serious Adverse Events (participants affected / at risk) | 1/3 | 5/22 | 1/6 | 1/4
Other Adverse Events (participants affected / at risk) | 3/3 | 22/22 | 6/6 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 5mg (N=3) | Expansion (N=22) | Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 6mg (N=6) | Fulvestrant 500mg, Palbociclib 125mg and Erdafitinib 8mg (N=4)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 5mg (N=3) | Expansion (N=22) | Fulvestrant 500mg/Palbociclib 125mg/Erdafitinib 6mg (N=6) | Fulvestrant 500mg, Palbociclib 125mg and Erdafitinib 8mg (N=4)
Oral mucositis (Gastrointestinal disorders) | 3 (10) | 13 (22) | 5 (11) | 3 (8)
Constipation (Gastrointestinal disorders) | 3 (3) | 14 (23) | 2 (3) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 12 (14) | 4 (4) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 10 (20) | 3 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (4) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 2 (2) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Dyspesia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil decreased (Investigations) | 3 (7) | 15 (35) | 4 (5) | 1 (2)
White blood cell decreased (Gastrointestinal disorders) | 3 (6) | 11 (19) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 1 (3) | 9 (11) | 2 (4) | 0 (0)
Alkaline phosphatase increased (Investigations) | 2 (3) | 2 (2) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 3 (6) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 1 (3)
Creatinine increased (Investigations) | 1 (1) | 3 (5) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (4) | 2 (3) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 2 (3) | 12 (20) | 3 (6) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3) | 11 (13) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (7) | 4 (5) | 2 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (10) | 0 (0) | 0 (0)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-paular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (7) | 12 (13) | 4 (4) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 4 (7) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (3)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (3) | 12 (24) | 5 (8) | 1 (1)
Pain (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Limb edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglyemia (Metabolism and nutrition disorders) | 2 (4) | 6 (7) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (5) | 3 (4) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (7) | 3 (3) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 3 (11) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eyes (Eye disorders) | 1 (1) | 9 (10) | 2 (2) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (11) | 7 (11) | 2 (6) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3) | 4 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperparathyroidism (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/96/NCT03238196/Prot_SAP_000.pdf